CLINICAL TRIAL: NCT00004910
Title: A Pilot Phase I/II Trial of Enteral Wallstents for Duodenal Obstruction in the Setting of Malignancy
Brief Title: Endoscopic Placement of Metal Stents in Treating Patients With Cancer- Related Duodenal Obstruction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Supportive Care
Other Study IDs: NU 98CC2; NU-98CC2; NCI-G00-1703
Record Dates: First submitted 2000-03-07; First posted 2003-05-09 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-05

CONDITIONS: Colorectal Cancer; Constipation, Impaction, and Bowel Obstruction; Extrahepatic Bile Duct Cancer; Gastric Cancer; Gastrointestinal Carcinoid Tumor; Gastrointestinal Stromal Tumor; Pancreatic Cancer; Quality of Life; Small Intestine Cancer
Keywords: stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; stage I gastric cancer; stage II gastric cancer; stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer; stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; recurrent pancreatic cancer; recurrent colon cancer; localized gastrointestinal carcinoid tumor; regional gastrointestinal carcinoid tumor; metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; small intestine adenocarcinoma; small intestine lymphoma; small intestine leiomyosarcoma; localized extrahepatic bile duct cancer; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; recurrent small intestine cancer; constipation, impaction, and bowel obstruction; quality of life; gastrointestinal stromal tumor; stage IV pancreatic cancer
MeSH Terms: conditions — Colorectal Neoplasms; Constipation; Intestinal Obstruction; Bile Duct Neoplasms; Stomach Neoplasms; Gastrointestinal Stromal Tumors; Pancreatic Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: bowel obstruction management
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: The use of endoscopy to place metal stents in the duodenum is less invasive than surgery for treating cancer-related duodenal obstruction and may have fewer side effects and improve recovery.

PURPOSE: Phase I/II trial to study the effectiveness of endoscopic placement of metal stents in treating patients who have cancer-related obstruction of the duodenum.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response and clinical outcome in patients with duodenal obstruction secondary to malignancy treated with enteral Wallstents.
* Evaluate the efficacy and safety of this treatment in these patients.
* Evaluate the quality of life of these patients after enteral Wallstent placement.

OUTLINE: Patients undergo enteral Wallstent placement through an endoscope under fluoroscopic guidance into the duodenum.

Quality of life is assessed at 48 hours and 6 months after procedure.

Patients are followed at 48 hours, 30 days, 6 months, and then yearly thereafter until death.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Endoscopically confirmed localized tumor as the cause of duodenal obstruction

  * All primary tumor types are eligible
* No prior duodenal Wallstents
* Must have symptoms of gastrointestinal obstruction, including:

  * Inability to move bowels, absence of flatus, nausea/vomiting, abdominal pain, or diarrhea

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-3

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count greater than 50,000/mm^3

Hepatic:

* INR no greater than 1.5 times upper limit of normal

Renal:

* Not specified

Cardiovascular:

* No cardiac condition

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No significant active infection (e.g., pneumonia, peritonitis, or wound abscess) that would preclude endoscopy
* No other serious concurrent illness
* No uncontrolled metabolic disease (e.g., diabetes mellitus or hypothyroidism)
* No dementia, psychiatric disorder, or altered mental status that would preclude compliance
* History of other neoplastic disease allowed
* Veterans Administration patients are not eligible

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Prior or concurrent chemotherapy allowed

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior or concurrent radiotherapy allowed

Surgery:

* At least 3 weeks since prior surgery and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-01; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Willis G. Parsons, MD, PC, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States